CLINICAL TRIAL: NCT06633991
Title: Expectancies About Positive Outcomes and Their Possible Potentiating Role of Standard Treatment in Migraine Patients
Brief Title: Expectancies in Migraine Patients
Acronym: EXPMIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Fiammetta Cosci, Professor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXPMI
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Migraine
Keywords: expectations; placebo effect; migraine; verbal instrucitons
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: control vs experiemntal condition
Who Masked: Participant
Masking Description: participants did not know whether they were allocated to the control or the experimental condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instructions inducing hope and optimism (Experimental): The verbal instruction inducing more hope and optimism will be: "The present therapy is a very effective one for your specific type of headache. By taking it, a large number of patients experienced significant pain relieve and improvement in functional capacity
  Interventions: Procedure: verbal instructions
- neutral instructions (Placebo Comparator): The verbal instruction inducing hope and optimism will be: "The present therapy is an effective one for your specific type of headache. By taking it, a large number of patients experienced pain relieve and improvement in functional capacity".
  Interventions: Procedure: verbal instructions

INTERVENTIONS:
Procedure: verbal instructions — verbal instructions inducing hope and optimism were administered as experimental condition vs neutral instructions (i.e., instructions not able to induce hope and optimism although realistic ones)
  Other Names: verbal instrucitons

SUMMARY:
The aim of the present study is to examine whether the standard treatment prescribed to migraine patients is potentiated when coupled with a verbal instruction inducing more hope and optimism. In order to achieve the goal, outpatients with low-frequency episodic migraine diagnoses (<8 attacks per month) and outpatients with chronic migraine diagnoses (>15 attacks per month) will be screened and enrolled, thereafter they will be exposed to verbal instruction inducing more hope and optimism or to verbal instruction inducing hope and optimism together with standard treatment. We hypothesize that the group receiving verbal instruction inducing more hope and optimism would develop larger improvements in all outcome measures.

DETAILED DESCRIPTION:
Study design and sample Cohort study with longitudinal detection of the endpoints of interest for the study (See section "Instruments").

Among the new patients or outpatients already assisted at the SOD Center Headache and Clinical Pharmacology of the University Hospital (AOU) Careggi, the candidates eligible for participation will be identified according to the inclusion and exclusion criteria listed below and participation will be proposed. Patients who, after being informed will consent through explicit and written informed consent to participate in the study, will be enrolled. A total of 100 subjects will be enrolled. Each participant will be able to withdraw the consent for participation at any time without providing justification. The request will invariably be accepted, and the subject's data will be excluded from the study.

Inclusion criteria for cases:

1. Incident or prevalent diagnosis of low-frequency episodic migraine or chronic migraine according to ICHD criteria version 3 beta 2013.
2. Age of at least 18 years.
3. Signature of informed consent.

Exclusion criteria for cases:

1. Standard treatment proposed different from topiramate, amitriptyline, valproate, β-blockers.
2. Inability to understand and want.

Procedure Migraine patients will receive a baseline assessment aimed at formulating or confirming the diagnosis of migraine based on a specific set of questions that doctors of the SOD Center of Headache and Clinical Pharmacology use routinely. The doctors of the SOD Center of Headache and Clinical Pharmacology will inform migraine patients about the purposes and procedures of the study and will gather consent to participate in the study by them. Consent will be explicitly issued by signing a specific form. Thereafter, a psychologist will collect socio-demographic information, information relating to the pharmacological and non-pharmacological treatment in progress, information relating to the history of organic disease, based on a set of questions already used in the past. The interview will take about 30 minutes. Then, doctors of the SOD Center of Headache and Clinical Pharmacology will formulate the standard prescription based on their routine practice. Such prescription will be coupled to a verbal instruction inducing more hope and optimism or to a verbal instruction inducing hope and optimism, according to a random assignment. Block randomization of size two will be used. The allocation schedule will be created centrally by an independent researcher using a computerized random number generator; the other investigators will be blinded to the schedule.

The entire study will last 12 months. Each subject will be assessed before starting the treatment (i.e., baseline) and at 7-day, 15-day, 1-month, 2-month and 3-month follow-ups. Each subject will be asked to devote about two hours to the participation to the present study.

Instruments Socio-demographic information, information regarding pharmacological and non-pharmacological treatment and information concerning the clinical history of organic pathology will be collected through a special set of questions already used in the past. Participant data will be archived and processed only after appropriate anonymization. Each subject will receive an alphanumeric code which will be the only identification code on the questionnaires. The doctors of the SOD Center of Headache and Clinical Pharmacology will keep the documents in a special archive that will allow each patient to be associated with their own alphanumeric identification code. This document will allow the possible deletion of a patient's data, if the patient makes an explicit request.

Psychological variables will be measured using the following tools:

* Headache Impact Test (HIT-6): this 6-item instrument was designed to provide a global measure of adverse headache and migraine impact on patients' everyday life. It is intended for use in screening and monitoring patients with headaches in both clinical practice and clinical research. It includes 6 items measuring the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning, psychological distress and the severity of headache pain. The scoring ranges from 36 to 78, with a cutoff score of 50. The patient is asked to indicate the impact of headache in the past 4 weeks on a 6-point scale (never, rarely, sometimes, very often, always). Higher scores indicate a greater impact on the patient's life.
* A Numeric Rating Scale (NRS) assessing the intensity of migraine pain on a 11-point NRS (0 = no pain, 10 = worst imaginable pain) during the last migraine attack.
* Assessment of expectancies about the effects of the treatment on migraine. Before starting the treatment prescribed, the patient's expectancies of the reduction in migraine pain related to the treatment will be assessed asking the question "Based on the intensity of migraine pain during the last migraine attack, what intensity do you expect one week after the beginning of the new treatment?". The answer will be based on an 11-point NRS (0 = no pain, 10 = worst migraine pain). Expectancy will be computed as a difference value between the migraine pain of the last attack and the expected intensity in migraine pain one week after the beginning of the treatment. Negative mean values will indicate that pain reduction is expected. Positive values will indicate an expected increase in pain.

The above instruments will be administered immediately before starting the drug treatment, at 7 days, 15 days, 1 month, 2 months, 3 months.

In addition, at 7 days, 15 days, 1 month, 2 months, 3-month follow-ups, the Kellner's scale of change after treatment will be administered. This is a 9-point NRS (9 = much worse; 1 = much improved) assessing the level of change of migraine pain over the time.

Instructions The verbal instruction inducing more hope and optimism will be: "The present therapy is a very effective one for your specific type of headache. By taking it, a large number of patients experienced significant pain relieve and improvement in functional capacity The verbal instruction inducing hope and optimism will be: "The present therapy is an effective one for your specific type of headache. By taking it, a large number of patients experienced pain relieve and improvement in functional capacity".

The instruction will be given at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Incident or prevalent diagnosis of low-frequency episodic migraine or chronic migraine according to ICHD criteria version 3 beta 2013.
* Age of at least 18 years.
* Signature of informed consent.

Exclusion Criteria:

* Standard treatment proposed different from topiramate, amitriptyline, valproate, β-blockers.
* Inability to understand and want.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test | baseline, 7-day, 15-day, 1- and 3-month follow-ups
  self-report scale assessing the disability due to migraine
Intensity of migraine | baseline, 7-day, 15-day, 1- and 3-month follow-ups
  A Numeric Rating Scale (NRS) assessing the intensity of migraine pain on a 11-point NRS (0 = no pain, 10 = worst imaginable pain) during the last migraine attack

SECONDARY OUTCOMES:
Expectancies | baseline, 7-day, 15-day, 1- and 3-month follow-ups
  Assessment of expectancies about the effects of the treatment on migraine. Before starting the treatment prescribed, the patient's expectancies of the reduction in migraine pain related to the treatment will be assessed asking the question "Based on the intensity of migraine pain during the last migraine attack, what intensity do you expect one week after the beginning of the new treatment?". The answer will be based on an 11-point NRS (0 = no pain, 10 = worst migraine pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Fiammetta COSCI, Florence, Italy

IPD SHARING:
Plan to Share IPD: No
IPD were made available only to the researchers directly involved in the data collection.